CLINICAL TRIAL: NCT00357396
Title: A Phase II Trial of a Chemotherapy Based Regimen of Intravenous Busulfan (Busulfex), Melphalan and Thiotepa as Myeloablative Regimen Followed by a T- Cell Depleted Allogeneic Hematopoietic Stem Cell Transplant From and HLA-Compatible Donor in the Treatment of High Risk Ewing's Sarcoma Family Tumors
Brief Title: Busulfan, Melphalan, and Thiotepa Followed By a Donor Stem Cell Transplant in Treating Patients With High-Risk Ewing's Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-059; MSKCC-05059
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-10

CONDITIONS: Sarcoma
Keywords: metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Therapeutics; Busulfan; Melphalan; Thiotepa; Peripheral Blood Stem Cell Transplantation

ARMS (1):
- Chemo followed by DSCT (Experimental): * Myeloablative preparative regimen: Patients receive busulfan IV over 2 hours every 6 hours on days -8 to -6, melphalan IV over 20 minutes on days -5 to -3, and thiotepa IV over 4 hours on day -2.
  * Allogeneic hematopoietic stem cell transplant: Patients undergo allogeneic bone marrow or T-cell depleted peripheral blood stem cell transplantation on day 0.
  * Graft-vs-host disease (GVHD) prophylaxis: Patients receive treatment according to institutional guidelines and are given treatment against infection.
  After completion of study treatment, patients are followed periodically for at least 3 years.
  Interventions: Biological: graft versus host disease prophylaxis/therapy; Drug: busulfan; Drug: melphalan; Drug: thiotepa; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: graft versus host disease prophylaxis/therapy
Drug: busulfan
Drug: melphalan
Drug: thiotepa
Procedure: allogeneic bone marrow transplantation
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy drugs, such as busulfan, melphalan, and thiotepa, before a donor stem cell transplant helps stop the growth of tumor cells and prepares the patient's bone marrow for the stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal tissues. Giving tacrolimus, sirolimus, and mycophenolate mofetil may stop this from happening.

PURPOSE: This phase II trial is studying how well giving busulfan together with melphalan and thiotepa followed by a donor stem cell transplant works in treating patients with high-risk Ewing's tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate disease-free and overall survival of patients with high-risk tumors of the Ewing's family treated with unmodified T-cell depleted allogeneic hematopoietic stem cell transplantation after cytoreduction comprising busulfan, melphalan, and thiotepa.
* Determine the regimen-related morbidity and mortality in these patients.
* Determine the incidence of acute and chronic graft-vs-host disease in patients treated with this regimen.
* Determine the biologic response of minimal residual disease in patients treated with this regimen.

OUTLINE: This is a prospective study.

* Myeloablative preparative regimen: Patients receive busulfan IV over 2 hours every 6 hours on days -8 to -6, melphalan IV over 20 minutes on days -5 to -3, and thiotepa IV over 4 hours on day -2.
* Allogeneic hematopoietic stem cell transplant: Patients undergo allogeneic bone marrow or T-cell depleted peripheral blood stem cell transplantation on day 0.
* Graft-vs-host disease (GVHD) prophylaxis: Patients receive treatment according to institutional guidelines and are given treatment against infection.

After completion of study treatment, patients are followed periodically for at least 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of high-risk tumors of the Ewing's family as defined by 1 of the following:

  * Biopsy-proven disease with distant metastases to sites other than the lung
  * Relapsed disease after completion of prior standard front-line therapy or high-dose chemotherapy
* Currently in complete remission (CR) with no evidence of disease (with or without minimal residual disease) or very good partial remission (i.e., CR with an abnormal bone scan) after prior standard or high-dose chemotherapy with local control
* HLA-compatible stem cell donor available

  * Compatible donors include those matched at both HLA-A, -B, -C, -DR and 1 of 2 -DQ alleles by high-resolution molecular typing
  * Related or unrelated donor

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 70-100% (≥ 16 years old) OR Lansky PS 70-100% (< 16 years old)
* LVEF > 50% at rest
* SGOT < 3 times upper limit of normal
* Bilirubin < 2.0 mg/dL (unless liver is involved with disease)
* Creatinine normal AND/OR creatinine clearance > 60 mL/min
* Lung diffusion capacity > 50% of predicted (corrected for hemoglobin) OR asymptomatic with a room air oxygen saturation of ≥ 98%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active uncontrolled viral, bacterial, or fungal infection
* No HIV-1 or -2 positivity

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior therapy with 100 mg/m² of melphalan
* No prior high-dose chemotherapy requiring autologous stem cell rescue
* No prior radiotherapy to > 50% of the pelvic marrow space

Max Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2005-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Prockop, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With HIGH RISK EWING'S SARCOMA FAMILY TUMOR: MELPHALAN & THIOTEPA TREATMENT OF HIGH RISK EWING'S SARCOMA FAMILY TUMOR
- Related Donors: Any consenting healthy family donor who is HLA compatible with the recipient will be considered as a potential donor for transplant
Period: Overall Study
Arm/Group | Patients With HIGH RISK EWING'S SARCOMA FAMILY TUMOR | Related Donors
Started | 6 | 4
Completed | 5 | 4
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With HIGH RISK EWING'S SARCOMA FAMILY TUMOR | Related Donors | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 1 | 4
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Patients With HIGH RISK EWING'S SARCOMA FAMILY TUMOR
Number analyzed (Participants) | 5
participants
  Very Good Partial Response (VGPR) | 4
  Complete Response (CR) | 1

ADVERSE EVENTS:
Arm/Group | Patients With HIGH RISK EWING'S SARCOMA FAMILY TUMOR | Related Donors
Serious Adverse Events (participants affected / at risk) | 4/6 | 0/4
Other Adverse Events (participants affected / at risk) | 6/6 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With HIGH RISK EWING'S SARCOMA FAMILY TUMOR (N=6) | Related Donors (N=4)
Constitutional Symptoms, other (General disorders) | 1 (1) | 0 (0)
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Infection w/ Gr 3/4 neut, Abdomen NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection w/ Gr 3/4 neut, Blood (Infections and infestations) | 1 (1) | 0 (0)
Liver dysfunction/failure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With HIGH RISK EWING'S SARCOMA FAMILY TUMOR (N=6) | Related Donors (N=4)
ALT, SGPT (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
AST, SGOT (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Alkaline phosphatase (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Amylase (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Cholesterol,high(hypercholestremia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Dermatology/Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal, other (Gastrointestinal disorders) | 3 (3) | 0 (0)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Hemorrhage, Urinary NOS (Renal and urinary disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Lipase (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Magnesium, high (hypermagnesemia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Magnesium, low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Mucositis (Clin exam)- Oral cavity (General disorders) | 2 (2) | 0 (0)
Nausea (General disorders) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
PTT (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Pain - Abdomen NOS (General disorders) | 1 (1) | 0 (0)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 4 (5) | 0 (0)
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Sodium, high (hypernatremia) (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Trglycrde, high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Vomiting (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes